CLINICAL TRIAL: NCT04589156
Title: Recurrent Acute Myocarditis : Characteristics, Etiology, Prognosis and Genetic Basis.
Brief Title: Recurrent Acute Myocarditis Registry
Acronym: RAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Rythmo20200818
Record Dates: First submitted 2020-08-31; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Myocarditis; Cardiomyopathy
Keywords: Recurrent acute myocarditis; Myocardial inflammation; Arrhythmogenic cardiomyopathy
MeSH Terms: conditions — Myocarditis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association between myocardial inflammation (clinically represented by acute myocarditis episodes) and the later development of an arrhythmogenic cardiomyopathy is widely elusive.

DETAILED DESCRIPTION:
Acute myocarditis (AM) is an inflammatory disease of the myocardium caused by different infectious and non-infectious triggers. It is a major cause of sudden cardiac death, with also long-term adverse outcomes in survivors. The incidence and predictive factors of recurrent AM (RAM) are unknown.

Arrhythmogenic cardiomyopathy (ACM) is a genetically-determined or acquired arrhythmogenic disorder of the myocardium. With an incidence of 1/5000, genetic ACM is the consequence of pathogenic variants in genes encoding for desmosomal and cytoskeleton proteins. Originally described as a right ventricular disease (ARVC), genetic ACM is increasingly recognized as a left (ALVC) or biventricular entity. Genetic ACM may manifest with various clinical presentations, with a predisposition to acute and chronic heart failure, ventricular arrhythmias and sudden cardiac death. Pathophysiology of genetic ACM at early stages remain widely elusive.

Myocardial inflammation has been consistently reported in patients with genetic ACM, but the exact nature of their association is a matter of debate. The temporal association between RAM episodes and the later diagnosis of genetic ACM is speculative, and it has been hypothesized recently that RAM episodes might reflect early active phases in the development of a genetic ACM.

The investigators aim to study the temporal association between RAM episodes and the later diagnosis of an ACM.

Consecutive patients with at least two episodes of AM and referred to a tertiary university referral center (pop. 1.500.000 inhabitants) for clinical expertise, follow-up and etiological work-out were prospectively included in this registry.

ELIGIBILITY:
Inclusion Criteria: patients with at least two episodes of acute myocarditis as defined by the European Society of Cardiology diagnostic criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with recurrent acute myocarditis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Sustained ventricular arrhythmia | 0 - 1 year after last acute myocarditis episode
  Any ventricular arrhythmia (VT/VF) :
  * sustained (lasting more than 30 seconds)
  * symptomatic or not (including sudden cardiac arrest)
  * induced or not (including during stress ECG, pharmacological challenge or electrophysiological study)
Genetic mutation | 0 - 1 year after last acute myocarditis episode
  Any genetic mutation (cardiomyopathy panel)

SECONDARY OUTCOMES:
Myocardial substrate characterization | 0 - 1 year after last acute myocarditis episode
  Cardiac magnetic resonance imaging (left and right ventricular ejection fractions, volumes, late gadolinium enhancement)
Nonsustained ventricular arrhythmia | 0 - 1 year after last acute myocarditis episode
  Any ventricular arrhythmia (VT/VF) :
  * nonsustained (lasting less than 30 seconds)
  * symptomatic or not
  * induced or not (including during stress ECG, pharmacological challenge or electrophysiological study)

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burke AP, Farb A, Tashko G, Virmani R. Arrhythmogenic right ventricular cardiomyopathy and fatty replacement of the right ventricular myocardium: are they different diseases? Circulation. 1998 Apr 28;97(16):1571-80. doi: 10.1161/01.cir.97.16.1571. PMID 9593562
- [Background] Bauce B, Basso C, Rampazzo A, Beffagna G, Daliento L, Frigo G, Malacrida S, Settimo L, Danieli G, Thiene G, Nava A. Clinical profile of four families with arrhythmogenic right ventricular cardiomyopathy caused by dominant desmoplakin mutations. Eur Heart J. 2005 Aug;26(16):1666-75. doi: 10.1093/eurheartj/ehi341. Epub 2005 Jun 7. PMID 15941723
- [Background] Bowles NE, Ni J, Marcus F, Towbin JA. The detection of cardiotropic viruses in the myocardium of patients with arrhythmogenic right ventricular dysplasia/cardiomyopathy. J Am Coll Cardiol. 2002 Mar 6;39(5):892-5. doi: 10.1016/s0735-1097(02)01688-1. PMID 11869858
- [Background] Chimenti C, Pieroni M, Maseri A, Frustaci A. Histologic findings in patients with clinical and instrumental diagnosis of sporadic arrhythmogenic right ventricular dysplasia. J Am Coll Cardiol. 2004 Jun 16;43(12):2305-13. doi: 10.1016/j.jacc.2003.12.056. PMID 15193698
- [Background] Asimaki A, Tandri H, Duffy ER, Winterfield JR, Mackey-Bojack S, Picken MM, Cooper LT, Wilber DJ, Marcus FI, Basso C, Thiene G, Tsatsopoulou A, Protonotarios N, Stevenson WG, McKenna WJ, Gautam S, Remick DG, Calkins H, Saffitz JE. Altered desmosomal proteins in granulomatous myocarditis and potential pathogenic links to arrhythmogenic right ventricular cardiomyopathy. Circ Arrhythm Electrophysiol. 2011 Oct;4(5):743-52. doi: 10.1161/CIRCEP.111.964890. Epub 2011 Aug 22. PMID 21859801
- [Background] Tanawuttiwat T, Sager SJ, Hare JM, Myerburg RJ. Myocarditis and ARVC/D: variants or mimics? Heart Rhythm. 2013 Oct;10(10):1544-8. doi: 10.1016/j.hrthm.2013.06.008. Epub 2013 Jun 14. No abstract available. PMID 23773988
- [Background] Protonotarios A, Wicks E, Ashworth M, Stephenson E, Guttmann O, Savvatis K, Sekhri N, Mohiddin SA, Syrris P, Menezes L, Elliott P. Prevalence of 18F-fluorodeoxyglucose positron emission tomography abnormalities in patients with arrhythmogenic right ventricular cardiomyopathy. Int J Cardiol. 2019 Jun 1;284:99-104. doi: 10.1016/j.ijcard.2018.10.083. Epub 2018 Oct 26. PMID 30409737
- [Background] Lopez-Ayala JM, Pastor-Quirante F, Gonzalez-Carrillo J, Lopez-Cuenca D, Sanchez-Munoz JJ, Oliva-Sandoval MJ, Gimeno JR. Genetics of myocarditis in arrhythmogenic right ventricular dysplasia. Heart Rhythm. 2015 Apr;12(4):766-73. doi: 10.1016/j.hrthm.2015.01.001. Epub 2015 Jan 20. PMID 25616123
- [Background] Martins D, Ovaert C, Khraiche D, Boddaert N, Bonnet D, Raimondi F. Myocardial inflammation detected by cardiac MRI in Arrhythmogenic right ventricular cardiomyopathy: A paediatric case series. Int J Cardiol. 2018 Nov 15;271:81-86. doi: 10.1016/j.ijcard.2018.05.116. Epub 2018 May 31. PMID 29885824
- [Background] Brown EE, McMilllan KN, Halushka MK, Ravekes WJ, Knight M, Crosson JE, Judge DP, Murphy AM. Genetic aetiologies should be considered in paediatric cases of acute heart failure presumed to be myocarditis. Cardiol Young. 2019 Jul;29(7):917-921. doi: 10.1017/S1047951119001124. Epub 2019 Jun 14. PMID 31198128
- [Background] Ader F, Surget E, Charron P, Redheuil A, Zouaghi A, Maltret A, Marijon E, Denjoy I, Hermida A, Fressart V, Gandjbakhch E. Inherited Cardiomyopathies Revealed by Clinically Suspected Myocarditis: Highlights From Genetic Testing. Circ Genom Precis Med. 2020 Aug;13(4):e002744. doi: 10.1161/CIRCGEN.119.002744. Epub 2020 Jun 10. No abstract available. PMID 32522011
- [Background] Piriou N, Marteau L, Kyndt F, Serfaty JM, Toquet C, Le Gloan L, Warin-Fresse K, Guijarro D, Le Tourneau T, Conan E, Thollet A, Probst V, Trochu JN. Familial screening in case of acute myocarditis reveals inherited arrhythmogenic left ventricular cardiomyopathies. ESC Heart Fail. 2020 Aug;7(4):1520-1533. doi: 10.1002/ehf2.12686. Epub 2020 May 1. PMID 32356610
- [Background] Caforio ALP, Re F, Avella A, Marcolongo R, Baratta P, Seguso M, Gallo N, Plebani M, Izquierdo-Bajo A, Cheng CY, Syrris P, Elliott PM, d'Amati G, Thiene G, Basso C, Gregori D, Iliceto S, Zachara E. Evidence From Family Studies for Autoimmunity in Arrhythmogenic Right Ventricular Cardiomyopathy: Associations of Circulating Anti-Heart and Anti-Intercalated Disk Autoantibodies With Disease Severity and Family History. Circulation. 2020 Apr 14;141(15):1238-1248. doi: 10.1161/CIRCULATIONAHA.119.043931. Epub 2020 Mar 2. PMID 32114801
- [Background] Belkaya S, Kontorovich AR, Byun M, Mulero-Navarro S, Bajolle F, Cobat A, Josowitz R, Itan Y, Quint R, Lorenzo L, Boucherit S, Stoven C, Di Filippo S, Abel L, Zhang SY, Bonnet D, Gelb BD, Casanova JL. Autosomal Recessive Cardiomyopathy Presenting as Acute Myocarditis. J Am Coll Cardiol. 2017 Apr 4;69(13):1653-1665. doi: 10.1016/j.jacc.2017.01.043. PMID 28359509
- [Background] Peretto G, Sala S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Campochiaro C, De Luca G, Foppoli L, Dagna L, Thiene G, Basso C, Della Bella P. Ventricular Arrhythmias in Myocarditis: Characterization and Relationships With Myocardial Inflammation. J Am Coll Cardiol. 2020 Mar 10;75(9):1046-1057. doi: 10.1016/j.jacc.2020.01.036. PMID 32138965
- [Background] Smith ED, Lakdawala NK, Papoutsidakis N, Aubert G, Mazzanti A, McCanta AC, Agarwal PP, Arscott P, Dellefave-Castillo LM, Vorovich EE, Nutakki K, Wilsbacher LD, Priori SG, Jacoby DL, McNally EM, Helms AS. Desmoplakin Cardiomyopathy, a Fibrotic and Inflammatory Form of Cardiomyopathy Distinct From Typical Dilated or Arrhythmogenic Right Ventricular Cardiomyopathy. Circulation. 2020 Jun 9;141(23):1872-1884. doi: 10.1161/CIRCULATIONAHA.119.044934. Epub 2020 May 6. PMID 32372669